CLINICAL TRIAL: NCT00200083
Title: SHAPE: Screened Health Assessment & Pacer Evaluation
Brief Title: Study of Weight Loss Using Gastric Stimulation in Obese Patients
Acronym: SHAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Medtronic Inc, Clinical research specialist
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 95-2002-015
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Obesity; Morbid Obesity
Keywords: Obesity; Morbid Obesity; SHAPE; IGS; Implantable Gastric Stimulator
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): All subjects enrolled will be implanted with an IGS system. The active group are those randomized to "on" and will receive active stimulation for 12 months.
  Interventions: Device: Transcend II Model 8848
- B (Placebo Comparator): All subjects enrolled will be implanted with an IGS system. The placebo group are those randomized to "off" and will receive no stimulation for 12 months.
  Interventions: Device: Transcend II Model 8848

INTERVENTIONS:
Device: Transcend II Model 8848 — All subjects will be implanted with the IGS device and then randomized to "on" or "off" for 12 months. After 12 months all subjects will be turned "on" through 24 month follow up.

SUMMARY:
The purpose of this study is to test the effect of an implanted device that stimulates the stomach to help obese patients lose weight.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate efficacy and safety of the IGS system in a population of patients with a BMI between 35 and 55 kg/m2.

SHAPE was a randomized, placebo-controlled, double-blind, multi-center pivotal study in which all subjects were implanted with the IGS system.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age at time of screening
* BMI of 35 to 55 kg/m2 at time of screening
* Patients with a reported history of five years of obesity (BMI > 30 kg/m2)

Exclusion Criteria:

* Patients who are excluded by the screening algorithm
* Patients scoring 29 or higher on the Binge Eating Scale Questionnaire
* Patients taking any weight loss medication or other drugs that can affect body weight

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2004-05; Primary Completion 2005-09 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Percent excess weight loss (%EWL) from baseline after 12 months from randomization. | Baseline, 12 months

SECONDARY OUTCOMES:
Percent excess weight loss (% EWL) from baseline at each study visit | Baseline and each study visit
Change from baseline in levels of satiety and appetite at each study visit. | Baseline and each study visit
Percentage change in body weight and BMI from baseline at each study visit | Baseline and each study visit
Proportion of subjects who attain ≥ 20% EWL from baseline after 12 months from randomization | Baseline and 12 months.
Proportion of subjects who lose ≥ 5% in body weight from baseline through Month 9, and maintain the weight loss for at least 3 months (i.e., through 12 months from randomization) | Baseline and each study visit.
Time to loss of weight maintenance or "relapse of weight loss" | Baseline and each study visit
Incidence of adverse events, Incidence of device complications, Change in blood chemistry and hematology laboratory assessments | During the course of the study until termination.

CONTACTS AND LOCATIONS:
Overall Officials: Obesity Study Team Obesity Study Team, Study Chair — Medtronic
Locations (8):
- United States (8):
  - Contact Medtronic for specific site information, Washington D.C., District of Columbia
  - Contact Medtronic for specfici site information, Gainsville, Florida
  - Contact Medtronic for specific site information, Chicago, Illinois
  - Contact Medtronic for specific site information, Boston, Massachusetts
  - Contact Medtronic for specific site information, Minneapolis, Minnesota
  - Contact Medtronic for specific site information, St Louis, Missouri
  - Contact Medtronic for specific site information, New York, New York
  - Contact Medtronic for specific site information, Philadelphia, Pennsylvania